CLINICAL TRIAL: NCT02025803
Title: A Phase 1, Open-Label, Non-randomized, Dose-Escalating Safety, Tolerability, and Pharmacokinetic Study of TAS-114 in Combination With Capecitabine in Patients With Advanced Solid Tumors
Brief Title: A Safety, Tolerability and Pharmacokinetic Study of TAS-114 in Combination With Capecitabine in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPU-TAS-114-101
Record Dates: First submitted 2013-12-27; First posted 2014-01-01 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Neoplasms
Keywords: Advanced solid tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAS-114/capecitabine (Experimental): See intervention description
  Interventions: Drug: TAS-114/capecitabine

INTERVENTIONS:
Drug: TAS-114/capecitabine — Part 1 (dose-escalation phase):
  Treatment cycles of TAS-114 and capecitabine orally BID for 14 days followed by 7 days rest until at least one of the discontinuation criteria are met TAS-114 dose starting at 20mg/m2/day with capecitabine dose of 760 mg/m2/day. TAS-114 doses will be escalated for each cohort up to 480mg/m2/day. If MTD is not reached by TAS-114 dose of 480mg/m2/day, the capecitabine dose will be escalated
  Part 2 (expansion phase):
  TAS-114 and capecitabine MTD established in Part 1 administered BID for 14 days followed by 7-day recovery period (21-day cycle).

SUMMARY:
The purpose of this exploratory study is to investigate the safety and determine the maximum tolerated dose (MTD) of TAS-114 in combination with capecitabine in patients with advanced solid tumors for which the patients have no available therapy likely to convey clinical benefit.

DETAILED DESCRIPTION:
In animal models, co-administration of TAS 114 and capecitabine has shown antitumor effects exceeding the maximum efficacy obtained by capecitabine alone. Developing a novel chemotherapy based on the combined use of TAS-114 and capecitabine may fulfill the need for more efficacious treatment for patients with advanced solid tumors.

The study, evaluating the safety, tolerability, pharmacokinetics, and preliminary antitumor activity of the TAS-114/ capecitabine regimen in patients with advanced solid tumors, will be conducted in two parts: a Dose-Escalation Phase (Part 1) to determine the MTD; and an Expansion Phase (Part 2) to further evaluate the safety and preliminary efficacy with the MTD.

ELIGIBILITY:
Inclusion Criteria:

1. Provided written consent
2. Is 18 years of age or older
3. Has histologically or cytologically confirmed advanced, measurable or non-measurable metastatic solid tumors for which the patients have no available therapy to convey clinical benefit Expansion Phase only: The target population should include at least

   1. 12 patients with breast cancer for whom 5 FU chemotherapy is the standard treatment
   2. 28 patients with refractory colorectal cancer.
4. May have received prior therapies for advanced or metastatic disease
5. Expansion Phase only: Has measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria (Version 1.1, 2009), ie, has at least one measurable lesion
6. Has ECOG performance status 0 or 1 on Cycle 1, Day 1
7. Is able to take medications orally
8. Has adequate organ function as defined by protocol
9. Women of childl-bearing potential must have a negative pregnancy test within 7 days prior to starting the study drug. Beth males and females must agree to adequate birth control if conception is possible during the study and for 6 months after the last dose
10. Is willing to and able to comply with scheduled visits and study procedures.

Exclusion Criteria:

1. Has a known DPD deficiency
2. Has had certain other recent treatment e.g. major surgery, anticancer therapy, extended field radiation, received investigational agent, within the specified time frames prior to study drug administration.
3. Certain serious illnesses or medical conditions
4. Is receiving concomitant treatment with drugs that may interact with capecitabine
5. Has had prior gastrectomy
6. Has known sensitivity to capecitabine or metabolites
7. Is a pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-11; Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
The MTD of TAS-114/ capecitabine (defined as the highest dose level at which less than 33% of the patients experience a Dose Limiting Toxicity (DLT) during the first cycle of treatment); DLTs defined by protocol | First cycle of treatment (ie. 21 days)
  Only drug-related toxicities during the first cycle are considered in the assessment of DLTs.

SECONDARY OUTCOMES:
Pharmacokinetic profiles (peak plasma concentration (Cmax) and area under the plasma concentration versus time curve (AUC) of TAS-114, capecitabine and it's metabolite 5-FU) | First cycle of treatment (ie. 21 days)
antitumor activity by tumor assessments according to RECIST criteria | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - IU Simon Cancer Center, Indianapolis, Indiana
  - Karmanos Cancer Institute, Detroit, Michigan